CLINICAL TRIAL: NCT02876081
Title: Phase II Study of Afatinib as Third- or Further-line Treatment for Patients With Stage IV Bronchial Adenocarcinoma, Harboring Wild-type EGFR, Expressing the Neurotensin - Neurotensin Receptor Complex
Acronym: THEN
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: medical decision
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Afatinib THEN
Record Dates: First submitted 2016-08-18; First posted 2016-08-23 (Estimated); Last update posted 2017-09-11 (Actual); Status verified 2017-09

CONDITIONS: SMALL CELL LUNG CARCINOMA
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — Afatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Afatinib — to evaluate the efficacy of afatinib, an EGFR TKI, on lung adenocarcinomas, EGFR wild-type, bearing the NTS/NTSR1 complex with a high level of expression

SUMMARY:
Lung cancer is the leading cause of cancer deaths in France, Europe and the world. 50% of lung cancers are of the adenocarcinoma subtype. 60% of patients present with a metastatic disease (stage IV) at the time of diagnosis. Approximately 10% of patients present with a mutation of the epidermal growth factor receptor (EGFR) requiring an EGFR tyrosine kinase inhibitor (EGFR-TKI), namely erlotinib, gefitinib or afatinib. For the majority of chemotherapy-naïve patients without addictive mutation, platinum-based chemotherapy, frequently the platinum - pemetrexed doublet, provides disease control rate of up to 70% and improves survival from approximately 4.5 with best supportive care alone to 15 months. However, patients with non-small cell lung cancer (NSCLC) usually relapse within 4 to 6 months and benefit from a second-line chemotherapy. Authorized drugs in this setting are pemetrexed, docetaxel and erlotinib. The prescription of erlotinib for unselected patients whose tumor does not harbor an EGFR mutation is questionable . In the second line setting, docetaxel provides less than 10% of partial responses and progression-free survival of 10 to 12 weeks. There are no standard options following failure of two previous lines of standard chemotherapy. In view of these modest results, new agents and therapeutic strategies are greatly needed for this patient population.

Neurotensin (NTS) is a 13 amino acids peptide, present and biologically active in the central nervous system and in periphery. At the peripheral level, NTS is released by the endocrine cells of the intestinal mucosa after meals and acts as an endocrine hormone involved in the postprandial regulation of the motor functions of the gastrointestinal tract. The effects of NTS are mediated by three subtypes of receptor: NTSR1 and NTSR2 exhibit high and low affinity for NTS, respectively, and belong to the family of G protein receptors; NTSR3 is a single transmembrane domain receptor. Exogenous activation of NTSR1 leads to cell proliferation, survival, mobility and invasion in cancer cells from diverse origin. These effects are the result from the activation of kinases and effectors, such as PKC, MAPK, FAK, RHO-GTPase, RAS and Src. The PKC activation may induce MAPK by direct stimulation of Raf-1, or by transactivation of the EGFR. The activation of MAPK via NTSR1 is mainly associated with uncontrolled cell growth. Both NTS and NTSR1 are expressed in 40% of lung tumors, whereas they are never expressed in the normal tissue. NTSR1 high expression is a negative prognostic factor in stage I to III operated lung adenocarcinomas. Sustained stimulation of NTSR1 results in the activation of MMP1, the release of EGF "like" ligands such as HB-EGF as well as neuregulin 1 NGR1 (a specific ligand for HER3) followed by EGFR, HER2 and HER3 overexpression and activation. Accordingly, xenografted tumors expressing NTS and NTSR1 show a positive response to erlotinib, whereas tumors void of NTSR1 expression have no detectable response.

Afatinib (BIBW2992) is a small molecule, selective and irreversible erbB family blocker. In preclinical models it effectively inhibits EGFR, HER2 and HER4 phosphorylation resulting in tumour growth inhibition and regression of established subcutaneous tumours derived from four human cell-lines known to co-express ErbB receptors.

Our claim is that patients harbouring the NTS/NTSR complex, without EGFR mutation, will respond to afatinib due to the sustained activation of EGFR/HER2 under neurotensin activation.

Presently, only EGFR mutated tumors are eligible to receive EGFR TKI representing 10% of all lung cancer patients. The aim of this study is to evaluate the efficacy of afatinib, an EGFR TKI, on lung adenocarcinomas, EGFR wild-type, bearing the NTS/NTSR1 complex with a high level of expression. This subpopulation of patients represents approximately 20% of lung adenocarcinomas.

ELIGIBILITY:
Inclusion Criteria:

* Patients with pathologic confirmation of EGFR wild type NSCLC Stage IV adenocarcinoma who have failed two lines of cytotoxic chemotherapy. One of the chemotherapy regimens must have been platinum-based.
* ECOG PS Score 0, 1
* Measurable disease according to RECIST version 1.1
* Life expectancy of at least 3 months.
* Written informed consent

Exclusion Criteria:

* Prior treatment with EGFR-targeting small molecules or antibodies.
* Radiotherapy or surgery (other than biopsy) within 4 weeks prior to randomisation.
* Active brain metastases (defined as stable for <4 weeks and/or symptomatic and/or requiring treatment with anticonvulsants or steroids and/or leptomeningeal disease).
* Known pre-existing interstitial lung disease.
* Significant or recent acute gastrointestinal disorders with diarrhoea as a major symptom e.g. Crohn's disease, malabsorption or CTC Grade ≥2 diarrhoea of any aetiology.
* History or presence of clinically relevant cardiovascular abnormalities such as uncontrolled hypertension, congestive heart failure NYHA classification of 3, unstable angina or poorly controlled arrhythmia. Myocardial infarction within 6 months prior to randomisation.
* Cardiac left ventricular function with resting ejection fraction of less than 50%.
* Any other concomitant serious illness or organ system dysfunction which in the opinion of the investigator would either compromise patient safety or interfere with the evaluation of the safety of the test drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2017-09-01 (Actual); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Assessment of disease-control rate | Two months after treatment
  disease-control rate with Complete Response CR, Partial response PR or Stable Disease S, after 2 months of treatment

SECONDARY OUTCOMES:
Assessment of Progression Free Survival PFS | Two months after treatment
Assessment of Overall Survival OS | Two months after treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Groupe Hospitalier Paris Saint Joseph, Paris, Île-de-France Region, France